CLINICAL TRIAL: NCT05755529
Title: Effects of Low LH Serum Levels on Oocyte Retrieval, Fertilization Rate and Embryo Quality During Controlled Ovarian Stimulation: Results From a Prospective Cohort Analysis
Brief Title: Effects of Low LH Serum Levels on Ovarian Pick-up Outcome
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Palermo (Other)
Responsible Party: Principal Investigator, Andrea Etrusco, Principal investigator, University of Palermo
Other Study IDs: LH-OS-1
Record Dates: First submitted 2023-02-08; First posted 2023-03-06 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2023-03

CONDITIONS: Infertility, Female; ART
Keywords: embryo quality; LH levels; Oocyte retrieval
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Luteinizing hormone (LH) plays a key role for normal follicular development and oocyte maturation in controlled ovarian stimulation. In particular, LH stimulates the proliferation and differentiation of theca cells for the secretion of androgens, which synergistically increase the production of estrogen. This study aimed to investigate the effects of low LH concentrations on oocyte retrieval, fertilization and embryo development in patients undergoing in vitro fertilization/intracytoplasmic sperm injection (IVF/ICSI). Patients undergoing IVF/ICSI were prospectively analyzed, subdividing them into three groups according to their age. Serum LH levels were evaluated at day 3, during stimulation (day 10) and before ovulation induction (day 12).

ELIGIBILITY:
Inclusion Criteria:

age between 18 and 40 years, body mass index 18-29 kg/m 2 , regular menstrual cycles, normal uterine cavity assess by hysteroscopy, normal uterus and ovaries at transvaginal sonography,

Exclusion Criteria:

abnormal cervical cytology, affected by any other endocrinological, metabolic, autoimmune, and gynecological disease.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women who received ovarian stimulation with follitropin alfa (Gonal F, Merck Serono, Germany) and ganirelix (Fyremaldel, Sun Pharma, Italy).
Sampling Method: Non-Probability Sample
Enrollment: 43 (Estimated)
Dates: Start 2023-03 (Estimated); Primary Completion 2023-03 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Oocyte retrieval | immediately after the intervention
  number of retrieved oocytes after controlled ovarian stimulation

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Dragotto, Biologist, Principal Investigator — Clinica del Mediterraneo - Ragusa; Giovanni Bracchitta, M.D., Study Director — Clinica del Mediterraneo - Ragusa; Antonio Simone Laganà, M.D., Ph.D., Study Chair — University of Palermo; Andrea Etrusco, M.D., Study Chair — University of Palermo